CLINICAL TRIAL: NCT06990620
Title: A Prospective, Multicenter, Single-Arm Study on the Efficacy and Safety of Transarterial Chemoembolization Combined With Ivonescimab in Unresectable, Non-Metastatic Hepatocellular Carcinoma
Brief Title: TACE Plus Ivonescimab for Unresectable Non-Metastatic HCC
Acronym: TACE HCC
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lunxiu Qin, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Huashan011
Record Dates: First submitted 2025-05-17; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE+AK112 (Experimental)
  Interventions: Combination Product: TACE+AK112

INTERVENTIONS:
Combination Product: TACE+AK112 — TACE+AK112 (PD-1/VEGF bi-antibody, 20mg/kg, ivgtt, Q3W)

SUMMARY:
This study is a single-arm, multicenter, prospective clinical trial designed to evaluate the efficacy and safety of Transarterial Chemoembolization (TACE) combined with envafolimab in patients with unresectable, non-metastatic hepatocellular carcinoma (HCC), while exploring potential biomarkers associated with treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, male or female
* Patients with histologically or pathologically confirmed hepatocellular carcinoma (HCC), or Patients meeting the clinical diagnostic criteria for hepatocellular carcinoma as defined by the American Association for the Study of Liver Diseases (AASLD)
* BCLC Intermediate (B) or Advanced (C) stage, with liver-confined disease and ineligible for curative options (e.g., resection, transplant, or ablation)
* Child-Pugh Class A (score 5-6) or Class B (score 7)
* ECOG PS ≤1
* Measurable disease per RECIST 1.1 criteria
* Life expectancy >12 weeks
* Adequate organ function meeting the following laboratory values: Hematological: Absolute neutrophil count (ANC) ≥1.5×10⁹/L Platelet count (PLT) ≥75×10⁹/L Hemoglobin (HGB) ≥90 g/L Hepatic: Total bilirubin (TBIL) ≤3× upper limit of normal (ULN) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤5×ULN Serum albumin ≥28 g/L Note: Patients may be enrolled if values stabilize after standard liver support therapy for ≥1 week, as assessed by the investigator. Renal: Serum creatinine (Cr) ≤1.5×ULN or Creatinine clearance ≥50 mL/min (calculated by Cockcroft-Gault formula) Coagulation: International normalized ratio (INR) ≤2×ULN or Activated partial thromboplastin time (APTT) ≤2×ULN
* Willing and able to provide written informed consent prior to any study-related procedures

Exclusion Criteria:

* Patients with histopathologically confirmed variant hepatocellular carcinoma (HCC) subtypes, including: Fibrolamellar hepatocellular carcinoma Sarcomatoid hepatocellular carcinoma Mixed hepatocellular-cholangiocarcinoma
* Prior local therapy targeting the index lesion(s), including but not limited to: Transarterial chemoembolization (TACE) Transarterial embolization (TAE) Transarterial radioembolization (TARE) Hepatic arterial infusion chemotherapy (HAIC) Radiofrequency ablation (RFA) Cryoablation High-intensity focused ultrasound (HIFU) Radiation therapy
* Prior systemic anti-cancer therapy for hepatocellular carcinoma, including but not limited to: Molecular targeted agents (e.g., tyrosine kinase inhibitors, anti-angiogenic drugs) Conventional chemotherapy Immunotherapy: Immune checkpoint inhibitors (e.g., PD-1/PD-L1/CTLA-4 inhibitors) Immune checkpoint agonists Cellular immunotherapy (e.g., CAR-T, NK cell therapy) Biological therapy: Cancer vaccines Cytokines (e.g., interferons, interleukins) Growth factor inhibitors
* Macrovascular invasion meeting either of the following criteria: Portal vein tumor thrombus (PVTT): Vp3: Tumor thrombus involving the first-order branches (left or right portal vein) Vp4: Tumor thrombus involving the main portal trunk or extending beyond Hepatic vein/inferior vena cava (IVC) tumor thrombus
* History of bleeding events within 6 months prior to initial treatment, including but not limited to: Acute hemorrhage from esophageal or gastric varices caused by portal hypertension AND/OR 6. Untreated or inadequately treated esophageal/gastric varices with high bleeding risk, as assessed by the investigator
* Clinically significant cardiovascular or cerebrovascular disease, including any of the following within 3 months prior to initial treatment: Congestive heart failure (NYHA Class ≥II) Myocardial infarction Cerebrovascular accident (stroke/TIA) Unstable arrhythmia Unstable angina OR 8. History of congenital long QT syndrome OR 9. Screening ECG showing QTc interval >500 ms (calculated by Fridericia's formula)
* Active autoimmune disease requiring systemic treatment (e.g., disease-modifying agents, corticosteroids, immunosuppressants) within 2 years prior to initial treatment, with the following exceptions: Non-systemic replacement therapies (e.g., thyroxine, insulin, or physiologic corticosteroid replacement for adrenal/pituitary insufficiency)
* Known HIV-positive status or history of active acquired immunodeficiency syndrome (AIDS)
* History of allogeneic stem cell transplantation or solid organ transplantation
* History of other active malignancies within 5 years prior to initial treatment, except for those with negligible risk of metastasis or death (e.g., 5-year overall survival rate >90%), including: Adequately treated carcinoma in situ of the cervix Non-melanoma skin cancer Localized prostate cancer (Gleason score ≤6, treated if required) Superficial bladder cancer (Ta/Tis, non-invasive)
* Women who are pregnant or breastfeeding
* Concurrent participation in another clinical trial, unless: It is a non-interventional study (e.g., observational/registry study), OR The patient is in the follow-up phase of an interventional trial, defined as: ≥4 weeks since last dose in the prior trial, OR ≥5 half-lives of the investigational drug (whichever is shorter)
* Systemic corticosteroid (>10 mg/day prednisone or equivalent) or other immunosuppressive therapy within 2 weeks prior to initial treatment, with the following exceptions: Adrenal replacement therapy (prednisone ≤10 mg/day or equivalent) Topical, ocular, intra-articular, intranasal, or inhaled corticosteroids with minimal systemic absorption Short-term corticosteroid prophylaxis for hypersensitivity reactions (e.g., premedication for CT scans)
* Any clinical or laboratory abnormality or compliance issue that, in the investigator's judgment, would preclude safe participation in the study
* Any condition that, in the investigator's opinion, may compromise patient safety or study integrity, including but not limited to: Clinically significant abnormal laboratory values not meeting specified thresholds Compliance concerns that may affect protocol adherence Other medical/psychosocial factors rendering the patient unsuitable for study participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Tumor assessments (per RECIST 1.1) every 6 weeks for the first 54 weeks relative to the date of randomization and then every 12 weeks thereafter. Assessed up to maximum of approximately 36 months.
  Disease assessments based on investigator assessments were determined by using RECIST version 1.1 guidelines. The ORR was defined as the percentage of patients with confirmed complete response (CR) or confirmed partial response (PR). The CR was defined as disappearance of all target and non-target lesions and no new lesions. The PR was defined as ≥ 30% decrease in the sum of diameters of target lesions (compared to baseline) and no new non-target lesion.